CLINICAL TRIAL: NCT00341666
Title: Regulation of Innate and Adaptive Immune Responses in Individuals Infected Concurrently With Malarial and Filarial Parasites
Brief Title: Immune Response Regulation in People Infected Concurrently With Malarial and Filarial Parasites
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906135; 06-I-N135
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-15

CONDITIONS: Malaria; Filarial Infection
Keywords: Immune Regulation; Co-Infection; Filariasis; Immunology; Filarial Infection
MeSH Terms: conditions — Malaria; Coinfection; Filariasis

SUMMARY:
This study, conducted by NIH and the University of Bamako in Mali, Africa, will study the effect of concurrent infections with malaria and filariasis on patients' immune response. Lymphatic filariasis is caused by infection with very small parasitic worms called Wuchereria bancrofti that are acquired from mosquitoes. The worms may cause no illness in many who are infected, but is some, they can cause swelling of the arms, legs, breast and genitalia, which may progress to permanent swelling referred to as elephantiasis. Malaria is caused by Plasmodium falciparum, another parasite that is spread by mosquitoes. It can cause fevers, headaches, body aches and weakness, and, if untreated, it can cause severe illness and death.

The 8-month study will analyze measures of immune function in blood cells from people with or without filarial infections who become infected with malaria. The goal of the studies is to see if having a filarial worm infection affects immunity against malaria. Results of analysis of immune function in persons with malaria but without filaria infections will be compared with those harboring both filaria and malaria infections and also with results from healthy control subjects.

Healthy individuals and patients with malaria and filarial infections between 1 and 8 years of age and between 18 to 65 years of age who live in N'Tessoni and healthy individuals living in Bamako, Mali (controls), may be eligible for this study.

Participants have blood samples collected as follows during the study:

* A blood sample will be collected at the beginning of the study. Individuals found to have the filarial worm infection have a second sample drawn at nighttime when the filarial worms are present in the blood. Treatment for filaria infection will be offered to all infected individuals at the end of the study.
* A second sample will be collected during malaria season. Subjects will be interviewed about their health during the malaria season and re-tested for filarial and malaria infections with a finger-prick test. Those who test positive for malaria will be offered treatment to begin immediately after collection of the donated blood sample..
* A third sample will be collected after the end of the malaria season. Subjects will be interviewed again about their health and re-tested for filarial and malaria infections with a finger prick test. Those who have positive results for either infection will be offered treatment after collec...

DETAILED DESCRIPTION:
Residents of malaria-endemic regions are frequently exposed to a variety of other parasites concurrently with malarial parasites. In Mali, lymphatic filariasis co-exists in several regions highly endemic for malaria. Because of the chronicity of filarial infections and an associated bias towards the development of an adaptive immune response dominated by Th2 cytokines, a pre-existing filarial infection has the potential to alter the immune response towards incoming malarial parasites, clearance of which are considered to be dependent on a robust Th1 response. Conversely, immune responses to filarial parasites may be modulated in the presence of malarial parasites. The goal of this study is to determine the effect of concurrent infections with malarial and filarial parasites on innate and adaptive immune responses to homologous and heterologous antigens. We will characterize the responses of peripheral blood mononuclear cells to antigens derived from both filarial (Wuchereria bancrofti) and malarial (Plasmodium falciparum) parasites in groups of individuals with or without filarial infections and follow them through a malaria transmission season, when they are repeatedly exposed to malarial parasites, to determine how co-infection with the filarial parasite affects the cellular and humoral responses to malarial and filarial antigens. These studies may provide the basis for modifying treatment strategies of mass treatment of malaria in regions co-endemic for lymphatic filariasis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 1-8 years or age 18-65 years.

Either resident of N'Tessoni (for active cohort) or resident of Bamako (for control cohort).

EXCLUSION CRITERIA:

Pregnancy (for the adult cohort).

Hemoglobin less than or equal to 8g/dl.

Symptoms of malaria with any level of parasitemia.

Recent history or clinical evidence of prostration, bleeding, respiratory distress, seizures, coma or obtundation, jaundice, inability to drink, persistent vomiting.

History of allergy to sulfa or pyrimethamine-sulfadoxine.

Plans to relocate outside the immediate village vicinity during the study period.

Clinical evidence of severe and/or chronic illness as determined by the examining physician.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2006-04-03; Study Completion 2011-07-15

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bamako, Faculty of Medicine, Pharmacy and Odontostomatology, Bamako, Mali

REFERENCES:
- [Background] Breman JG, Egan A, Keusch GT. The intolerable burden of malaria: a new look at the numbers. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):iv-vii. doi: 10.4269/ajtmh.2001.64.iv. No abstract available. PMID 11425185
- [Background] Gupta S, Snow RW, Donnelly CA, Marsh K, Newbold C. Immunity to non-cerebral severe malaria is acquired after one or two infections. Nat Med. 1999 Mar;5(3):340-3. doi: 10.1038/6560. PMID 10086393
- [Background] World Health Organization. Sixth meeting of the Technical Advisory Group on the Global Elimination of Lymphatic Filariasis, Geneva, Switzerland, 20-23 September 2005. Wkly Epidemiol Rec. 2005 Nov 18;80(46):401-8. No abstract available. English, French. PMID 16316047